CLINICAL TRIAL: NCT07150728
Title: The Effectiveness of Dignity Therapy in Terminal Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(I)-20220202
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2022-12

CONDITIONS: End of Life Patients
Keywords: End of life patients, dignity therapy, dignity, demoralization, depression
MeSH Terms: conditions — Depression | interventions — Dignity Therapy; Hospice and Palliative Care Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dignity therapy (Experimental): Dignity therapists use the "Dignity Psychotherapy Question Protocol" to guide patients through life's most important issues, providing them with the opportunity to participate in and discuss the things they would like their families to remember them for. During the process, dignity therapists use audio recording to fully record, transcribe, and edit the interview material, creating a valuable record that the patient wishes to preserve. The edited document is then returned to the patient, who then gives it to their family members.
  Interventions: Behavioral: dignity therapy
- Hospice palliative care (Placebo Comparator): Participants routinely performed hospice palliative care
  Interventions: Behavioral: Hospice palliative care

INTERVENTIONS:
Behavioral: dignity therapy — Dignity therapists use the "Dignity Psychotherapy Question Protocol" to guide patients through life's most important issues, providing them with the opportunity to participate in and discuss the things they would like their families to remember them for. During the process, dignity therapists use audio recording to fully record, transcribe, and edit the interview material, creating a valuable record that the patient wishes to preserve. The edited document is then returned to the patient, who then gives it to their family members.
  Arms: dignity therapy
Behavioral: Hospice palliative care — Participants regularly receive hospice care
  Arms: Hospice palliative care

SUMMARY:
Maintaining patient dignity is the moral obligation and an important ethical consideration of health professionals; it is also the primary connotation of medical care. Previous research revealed that terminal patients had moderate to severe dignity loss, and approximately 40% of them suffered from dignity-related distress, which required assistance from health professionals. This is a second- and third-year study project. The first-year study established and developed the localized "Terminal Patient Dignity Model" and "Terminal Patient Dignity Scale" for Taiwan. At present, the reliability and validity of the scale are being continuously tested. The second-year study adopts a longitudinal study design. The dignity therapy is referred for intervention. It adopts the randomized controlled experimental study method. Patients with terminal illness in a medical center will be randomly assigned to two groups, and each group is expected to have 34 patients. The experimental group will be provided with dignity therapy, whereas hospice palliative care will be adopted for the control group. Dignity, demoralization, depression, and other indicators will be measured in the pretest, immediately after the intervention, at 1 month and 3 months. In the third year, the study project will continue the intervention scheme and track the results of dignity, demoralization, depression, and other indicators at 6 and 9 months after the intervention. This study can help understand the status of dignity among terminal patients in Taiwan, and extend the terminal patient dignity scale and dignity therapy to noncancer terminal patients, in order to provide appropriate care to maintain dignity. It is also expected to provide a reference for the government to formulate empirical care policies on dignity therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with a terminal illness by their attending physician, whose disease has progressed to the point where death is inevitable, and who are receiving palliative care such as hospice care, hospice home care, or hospice co-care.
2. Patients aged 20 or above.
3. Patients who can communicate in Mandarin or Taiwanese.
4. Patients who are willing to participate in this research project and complete the consent form after the purpose and process of the research are explained.

Exclusion Criteria:

1. Those diagnosed by a physician with dementia, delirium, or other organic brain disease.
2. Those who are unconscious and incapable of acting.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Patient Dignity Inventory Mandarin Version (PDI-MV) | Before dignity therapy, immediately after intervention, 1 month, 3 months
Demoralization Scale-Mandarin Version (DS-MV) | Before dignity therapy, immediately after intervention, 1st month, 3rd month
Patient Health Questionnaire-9 (PHQ-9) | Before dignity therapy, immediately after intervention, 1st month, 3rd month

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No